CLINICAL TRIAL: NCT00312611
Title: Screened Health Assessment & Pacer Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 801287; G030194
Record Dates: First submitted 2005-09-01; First posted 2006-04-10 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Gastric pacing device; Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Device: Transcend II Implantable Gastric Stimulator (IGS), Model 8848

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of the Transneuronix IGS System in a population of patients with a BMI between 35 and 55.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate efficacy and safety of the Transneuronix IGS System in a population of patients with a BMI between 35 and 55. Initially, a maximum of 150 patients will be followed for 12 months in a randomized, placebo-controlled, double-blind, multi-center study to evaluate efficacy and safety of the IGS. All patients will be implanted with the IGS System and randomized to a control group (IGS OFF) or a treatment group (IGS ON). Both groups will follow a 500kcal/day-deficit diet (Appendix A) and participate in monthly support group meetings (Appendix E). The study will last for 24 months after randomization. The sponsor plans to submit a PreMarket Approval (PMA) application when all patients have completed 12 months of post-randomization follow-up. After 12 months from randomization, patients will continue to be followed monthly for another year, during which all patients will receive gastric electrical stimulation and the long-term efficacy and safety and maintenance of weight loss will be evaluated. After 24 months from randomization, all remaining patients will have the option to enter an extension study for an additional four years, during which the long-term efficacy and safety and maintenance of weight loss will continue to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1) Ability to give informed consent 2) 18 to 65 years of age at time of screening 3) BMI of 35 to 55 at time of screening 4) Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods. Acceptable birth control methods are limited to oral contraceptives, implants, diaphragms, IUDs, or condoms with or without spermicide, and voluntary abstinence. The method of birth control must be documented and verified at follow-up.

  5) Patients with a reported history of five years of obesity (BMI > 30) 6) Patients who require pharmacological therapy for psychological disorders, either at study entry or after implant, must obtain a letter from a licensed psychologist/psychiatrist justifying the use of the medication for psychological reasons only (Appendix D).

  7) Patients must agree to follow the dietary component of the protocol as outlined in Appendix A and attend monthly support group meetings (Appendix E).

  8) Patients must be geographically stable and reside within a 2-hour commute from the clinical site (as determined by the investigator or study coordinator) and be able and willing to travel to the clinical site for all follow-up visits and monthly support group meetings.

Exclusion Criteria:

* 1) Patients who are excluded by the screening algorithm18, 19, 22 (Appendix C) 2) Patients scoring 29 or higher on the Binge Eating Scale Questionnaire (Appendix F) 3) Patients will undergo a psychological evaluation by a licensed psychologist or psychiatrist (Appendix D). Patients who are substance abusers or are identified as having borderline personality, bipolar disorder, or any other disorder that would make them inappropriate candidates, in the opinion of the psychologist/psychiatrist.

  4) Pregnant or lactating females 5) Prior surgery of GI tract as therapy for obesity 6) Prior surgery on the stomach for any reason 7) Other electrical stimulation devices 8) Patients with known history or under treatment for ulcers 9) Patients with a clinically significant hiatal hernia 10) Patients with motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation 11) Patients taking any weight loss medication or other drugs that can affect body weight (e.g. mirtazapine, laxatives, systemic glucocorticoids, neuroleptic agents, progestational steroids) within three months prior to screening 12) Patients who require continuous therapy with known ulcerogenic medication (e.g., aspirin, non-steroidal anti-inflammatory agents, COX-2 inhibitors) 13) Patients with a history of cardiac arrhythmia or severe cardiac disease (NYHA class III or IV) 14) Type I diabetes and poorly controlled Type II diabetes as evidenced by an HbA1c level greater than 10%. Those patients with an HbA1c between 8% and 10% and who have ongoing symptoms of hyperglycemia, including unexplained weight loss or significant polyuria, polydipsia, or a fasting glucose level above 180 mg/dl* within 5 days prior to implantation, will be excluded.

  * If the fasting glucose level is above 180 mg/dl during screening, the patient will not be excluded from the study but be treated for hyperglycemia. Laboratory tests, including a fasting glucose level, will be repeated for all patients within 5 days prior to implantation.

  15) Any diabetic patients on non-steady treatment with thiazolidinediones (Actos or Avandia) within past three months prior to screening 16) Patients with a history of Barrett's esophagus 17) Patients who have severe weight-related co-morbid diseases that require immediate weight loss (e.g., life-threatening sleep apnea) 18) Patients with any serious health condition not related to their weight 19) Use of another investigational agent within 30 days prior to screening 20) Patients whom the investigator or study coordinator considers to be unable or unwilling to fulfill study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Percentage excess weight loss (%EWL) from baseline after 12 months from randomization
This study is designed to detect at least a mean 10% difference between the treatm

SECONDARY OUTCOMES:
% EWL from baseline at each study visit
% change in body weight (BW)and BMI from baseline at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: David Sarwer, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.medtronic.com